CLINICAL TRIAL: NCT03651869
Title: Mechanisms Linking Obsessive-Compulsive Symptoms and Tobacco Dependence
Brief Title: Effects of Nicotine in Tobacco Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Illinois Institute of Technology (Other)
Responsible Party: Principal Investigator, Adam Leventhal, Professor of Preventive Medicine and Psychology, Director of the Health, Emotion, and Addiction Laboratory, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 28IR-0063
Record Dates: First submitted 2018-08-23; First posted 2018-08-29 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Smoking, Tobacco; Smoking (Tobacco) Addiction
Keywords: Smoking
MeSH Terms: conditions — Tobacco Smoking; Smoking; Behavior, Addictive | interventions — Sugp2 protein, mouse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Condition 1 (Experimental)
  Interventions: Drug: Cigarette 1; Drug: Patch 1
- Condition 2 (Experimental)
  Interventions: Drug: Cigarette 2; Drug: Patch 1
- Condition 3 (Experimental)
  Interventions: Drug: Cigarette 1; Drug: Patch 2
- Condition 4 (Experimental)
  Interventions: Drug: Cigarette 2; Drug: Patch 2

INTERVENTIONS:
Drug: Cigarette 1 — Cigarette containing between 0mg nicotine and the conventional amount of nicotine (0.8mg)
  Arms: Condition 1; Condition 3
Drug: Cigarette 2 — Cigarette containing between 0mg nicotine and the conventional amount of nicotine (0.8mg)
  Arms: Condition 2; Condition 4
Drug: Patch 1 — A patch containing between 0mg nicotine and the conventional amount of nicotine (21mg)
  Arms: Condition 1; Condition 2
Drug: Patch 2 — A patch containing between 0mg nicotine and the conventional amount of nicotine (21mg)
  Arms: Condition 3; Condition 4

SUMMARY:
This study will examine mechanisms linking Obsessive-Compulsive Disorder symptomatology to tobacco dependence.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years old
* Daily smoking at least 2 years

Exclusion Criteria:

* Currently pregnant or breastfeeding.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Smoking Urge | Throughout study completion, an average of two weeks.
  Smoking urge is measured using questionnaires that ask about a desire to smoke.

CONTACTS AND LOCATIONS:
Overall Officials: Adam M Leventhal, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No